CLINICAL TRIAL: NCT02542345
Title: Comparative Assessment of Coronary MR Angiography Vs Coronary Multislice CT After Coronary Artery Reimplantation in Children and Young Adults.
Acronym: IRCADO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Collaborators: Hopital Universitaire Robert-Debre (Other); Amiens University Hospital (Other); University Hospital, Caen (Other); University Hospital, Rouen (Other); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00372-39
Record Dates: First submitted 2015-09-01; First posted 2015-09-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-03

CONDITIONS: Myocardial Ischemia
Keywords: Cardiac Multislice CT; MRI coronarography
MeSH Terms: conditions — Myocardial Ischemia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- magnetic resonance imaging (Experimental)
  Interventions: Procedure: magnetic resonance imaging

INTERVENTIONS:
Procedure: magnetic resonance imaging

SUMMARY:
This is a prospective, multicentric study conducted in order to evaluate if MRI coronarography is as powerful as Cardiac Multislice CT in detection of coronary abnormalities after coronary reimpantation in children over 5 yo, teenagers and young adults who underwent coronary reimplantation in childhood.

Newborns suffering from transposition of the great vessels who underwent at neonatal age an arterial switch operation (ASO) with coronary reimplantation, may develop in time with growth, stenosis, twist or elongation of the reimplanted coronary artery, which may cause myocardial ischemia. As well, aortic root surgery such as the Ross procedure and abnomalous coronary artery from pulmonary artery (ACAPA) reimplantation may lead to the same complications. Functional ischemic tests in a combination of three minimum are positive in only 75% of the cases . Silent ischemia due to coronary abnormality is to be detected in those patients.

In those patients, coronarography was recommended to be performed at least at 7 and 15 yo, without any clinical symptoms . It has also been recommended to examine those patients at 5, 10 and 15 yo as growth is the main cause for coronary abnormality development. Cardiac CT has been proven to be as efficient as coronarography to depict coronary reimplantation abnormalities .

Due to the invasiveness of angiography and to the development of cardiac CT, in our institution, the attitude is to performed cardiac CT instead of angiography with the same frequency in our patients.

Coronaro MRI has been established as a valid technique for evaluation of coronary arteries in patients after ASO .

The aim of this study is to evaluate if non contrast 3D MR coronarography is as powerful as Cardiac Multislice CT for the depiction of coronary anomalies.

All patients, with prior ASO, Ross or ACAPA reimplantation, refereed for cardiac CT and eligible for MRI, over 5yo are included in this prospective multi centric study.

Both examinations are performed on the same day after informed consent, from the patient or from both parents if minor.

Cardiac CT is performed according to the usual protocol in our institution, and MR coronaro angiography is performed as follow: excluding any contra indication to MR, the study requires one or two maximum 3D true FISP sequence without IV contrast injection, with cardiac gating, and free breathing.

3D images are evaluated blinded to the results of cardiac CT by two senior radiologists, with at least 5 years of experience in MR and CT cardiac imaging.

Comparison of the results is consolidated afterwards. Other elements evaluated are tolerance and feasibility of the examination.

The study is designed for four years and benefits from a grant from the Assistance Publique-Hopitaux de Paris.

ELIGIBILITY:
Inclusion Criteria:

* Non randomized patients requiring coronary imaging with cardiac CT
* for prior coronary reimplantation (arterial Switch, Ross procedure, ACAPA)
* aged of 5 years old or more,
* cooperating, requiring no sedation for MR examination
* Without contra indication to MR examination

Exclusion Criteria:

* Less than 5 years old
* Presenting a contra indication to MR examination
* Non cooperant
* Claustrophobic
* No informed consent
* For teenage girl, no pregnant test available

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-05 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of stenosis, performed on 3D workstations, reported in percentage (<50%, 50-70%, 70%) relative to the diameter of the normal vessel immediately below the stenosis. | The CT and MR examination are done the same day. There is no fixed time frame between the examinations and the measurements as the analysis is performed with a pooling of 30 patients at the same time. The time frame is variable, it ranges from 1 week to

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France